CLINICAL TRIAL: NCT01951287
Title: Impact of Fluid Milk on Post-meal Glycemia and Insulinemia in Overweight/Obese Adults With Normal or Impaired Glucose Tolerance or Type 2 Diabetes
Brief Title: Impact of Fluid Milk on Post-meal Glycemia and Insulinemia in Overwt/Obese Adults
Acronym: S37
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1303013430
Record Dates: First submitted 2013-09-12; First posted 2013-09-26 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Blood Glucose; Blood Insulin
MeSH Terms: interventions — Water; Economics; Milk

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Acute beverage (Water) consumption (Experimental): Acute beverage (Water)consumption with breakfast measuring blood glucose and insulin levels at specific time points. consumption with breakfast measuring blood glucose and insulin levels at specific time points.
  Interventions: Other: Acute beverage (water) consumption
- Acute beverage (Black Coffee) consumption (Experimental): Acute beverage (Black Coffee)consumption with breakfast measuring blood glucose and insulin levels at specific time points. consumption with breakfast measuring blood glucose and insulin levels at specific time points
  Interventions: Other: Acute beverage (Black Coffee) consumption
- Acute beverage (Orange Juice) consumption (Experimental): Acute beverage (Orange Juice)consumption with breakfast measuring blood glucose and insulin levels at specific time points. consumption with breakfast measuring blood glucose and insulin levels at specific time points
  Interventions: Other: Acute beverage (Orange Juice) consumption
- Acute beverage (Whole Milk) consumption (Experimental): Acute beverage (Whole Milk) consumption with breakfast measuring blood glucose and insulin levels at specific time points. consumption with breakfast measuring blood glucose and insulin levels at specific time points
  Interventions: Other: Acute beverage (Whole Milk) consumption
- Acute beverage (2% Milk) consumption (Experimental): Acute beverage (2% Milk) consumption with breakfast measuring blood glucose and insulin levels at specific time points. consumption with breakfast measuring blood glucose and insulin levels at specific time points
  Interventions: Other: Acute beverage (2% Milk) consumption
- Acute beverage (Skim Milk) consumption (Experimental): Acute beverage (Skim Milk)consumption with breakfast measuring blood glucose and insulin levels at specific time points. consumption with breakfast measuring blood glucose and insulin levels at specific time points
  Interventions: Other: Acute beverage (Skim Milk) consumption

INTERVENTIONS:
Other: Acute beverage (water) consumption — Acute beverage consumption includes water.
  Arms: Acute beverage (Water) consumption
Other: Acute beverage (Black Coffee) consumption — Acute beverage consumption includes black coffee.
  Arms: Acute beverage (Black Coffee) consumption
Other: Acute beverage (Orange Juice) consumption — Acute beverage consumption includes Orange Juice..
  Arms: Acute beverage (Orange Juice) consumption
Other: Acute beverage (Whole Milk) consumption — Acute beverage consumption includes whole milk
  Arms: Acute beverage (Whole Milk) consumption
Other: Acute beverage (2% Milk) consumption — Acute beverage consumption includes 2% milk
  Arms: Acute beverage (2% Milk) consumption
Other: Acute beverage (Skim Milk) consumption — Acute beverage consumption includes skim milk
  Arms: Acute beverage (Skim Milk) consumption

SUMMARY:
Blood sugar and insulin levels after a meal may be altered by the food and beverages a person consumes. Keeping a healthy blood sugar level may help prevent and manage type 2 diabetes and related diseases. This study will look at how drinking different common beverages (milk, low-fat milk, nonfat milk, orange juice, coffee, and water) with a meal changes blood sugar and insulin levels.

DETAILED DESCRIPTION:
The broad aim of the proposed research is to evaluate the effects of consuming milk and non-milk beverages with a breakfast meal on postprandial glucose and insulin responses in overweight and obese adults with varying levels of glucose tolerance (normal, pre-diabetic, type 2 diabetes). The investigators expect the consumption of fluid milk with breakfast to decrease the postprandial glucose response relative to other non-milk beverages (orange juice and sweetened coffee). Furthermore, the investigators expect that there will be no difference in the postprandial glucose or insulin response between varieties of fluid milk (skim, low-fat, and whole).

ELIGIBILITY:
Inclusion Criteria:

* 35-65 years old,
* BMI between 27-40 kg/m2,
* HbA1C less than 7.5%,
* weight stable (± 4.5 kg) for the previous 3 months
* willing to consume study foods and beverages.

Exclusion Criteria:

* using exogenous insulin,
* currently (or within the past 6 months) following a vigorous exercise regimen, or weight loss program,
* acute illness,
* smoking,
* pregnant or planning pregnancy in the next 3 months,
* lactose intolerant,
* weight changes of greater than ± 3 kg during the study period

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
plasma glucose levels | 6 mornings separated by at least a week, fasting and 30, 60, 60, 90, 120, 150,180,210,240 minutes postprandial
  Subjects will come to testing once a week for six weeks. Each testing day, subject will come in fasted, and a fasting blood draw will be taken. Subjects will then be fed a standard breakfast with one of the 6 beverages (coffee sweetened with sugar, orange juice, water, whole milk, skim milk, low fat milk). Blood will be taken at 30, 60, 60, 90, 120, 150,180,210,240 minutes after the meal.

SECONDARY OUTCOMES:
Plasma Insulin Levels | 6 mornings separated by at least a week, fasting and 30, 60, 60, 90, 120, 150,180,210,240 minutes postprandial
  Subjects will come to testing once a week for six weeks. Each testing day, subject will come in fasted, and a fasting blood draw will be taken. Subjects will then be fed a standard breakfast with one of the 6 beverages (coffee sweetened with sugar, orange juice, water, whole milk, skim milk, low fat milk). Blood will be taken at 30, 60, 60, 90, 120, 150,180,210,240 minutes after the meal.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Campbell, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States